CLINICAL TRIAL: NCT01753466
Title: The Water Intake Trial: Pilot Phase
Acronym: WIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Danone Global Research & Innovation Center (Industry)
Responsible Party: Principal Investigator, William Clark, Nephrologist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EAU-6607-GD
Record Dates: First submitted 2012-11-09; First posted 2012-12-20 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydration (Experimental): Participants who are randomized to the hydration-intervention group will be asked to consume 1.0 to 1.5 L water per day, depending on sex and weight, in addition to usual consumed beverages, for 6 weeks
  Interventions: Dietary Supplement: Hydration
- Control (No Intervention)

INTERVENTIONS:
Dietary Supplement: Hydration
  Arms: Hydration

SUMMARY:
The investigators are conducting a six-week randomized controlled pilot trial to assess the feasibility and safety of increased water intake in patients with chronic kidney disease.The investigators will study 30 patients (age 30 to 80 with an estimated glomerular filtration rate between 30 and 60 ml/min/1.73m2 and microalbuminuria [albumin to creatinine ratio >2.8 mg/mmol (if female) or >2.0 mg/mmol if male)].The investigators will randomize patients (in a 2:1 ratio) to a fluid-intervention group or control group. Participants who are randomized to the hydration-intervention group will be asked to consume 1.0 to 1.5 L water per day (depending on sex and weight) in addition to usual consumed beverages, for 6 weeks. Participants in the control group will be advised to consume their usual amount of fluid.

The investigators hypothesize that patients will be able to increase and maintain a higher fluid intake with stable blood chemistry, particularly serum sodium.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-80 years
* Able to provide informed consent and willing to complete follow-up visits.
* Estimated glomerular filtration rate between 30 and 60 ml/min/1.73m2
* Microalbuminuria [albumin to creatinine ratio >2.8 mg/mmol (if female) or >2.0 mg/mmol if male)]

Exclusion Criteria:

* Self-reported fluid intake >10 cups/day or 24-hr urine volume >3L.
* Enrolled in another randomized controlled trial that could influence the intervention, outcomes or data collection of this trial (or previously enrolled in this trial)
* Received one or more dialysis treatments in the past month
* Kidney transplant recipient (or on waiting list)
* Pregnant or breastfeeding
* History of kidney stones in past 5 years
* Less than two years life expectancy
* Serum sodium <130 mEq/L without suitable explanation
* Serum calcium >2.6 mmol/L without suitable explanation
* Currently taking hydrochlorothiazide >25 mg/d, indapamide >1.25 mg/d, furosemide >40 mg, or metolazone >2.5 mg/d
* Currently taking lithium
* Patient is under fluid restriction (< 1.5 L a day or more) for kidney disease, heart failure, or liver disease, AND meets any of the following criteria: i) end stage of the disease (heart left ventricular ejection fraction <40%, NYHA class 3 or 4, or end stage cirrhosis) or ii) hospitalization secondary to heart failure, ascites and/or anasarca

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
24-hour urine volume | 6 weeks (baseline and six weeks)
  Change in 24-hour urine volume between baseline and six weeks

CONTACTS AND LOCATIONS:
Overall Officials: William F Clark, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Derived] Sontrop JM, Huang SH, Garg AX, Moist L, House AA, Gallo K, Clark WF. Effect of increased water intake on plasma copeptin in patients with chronic kidney disease: results from a pilot randomised controlled trial. BMJ Open. 2015 Nov 24;5(11):e008634. doi: 10.1136/bmjopen-2015-008634. PMID 26603245
- [Derived] Clark WF, Sontrop JM, Huang SH, Gallo K, Moist L, House AA, Weir MA, Garg AX. The chronic kidney disease Water Intake Trial (WIT): results from the pilot randomised controlled trial. BMJ Open. 2013 Dec 20;3(12):e003666. doi: 10.1136/bmjopen-2013-003666. PMID 24362012